CLINICAL TRIAL: NCT06212505
Title: EVALUATION of the OVERALL HAEMOSTATIC CAPACITY of MIM8 with GLOBAL HAEMOSTASIS ASSAYS and FIBRIN CLOT ULTRASTRUCTURE
Acronym: Mim8-TGT
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_1202
Record Dates: First submitted 2024-01-08; First posted 2024-01-19 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Hemophilia a
Keywords: Mim8; TGT; Haemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The blood tubes required for this study will be taken during one of their visits and the 10 citrated tubes of 2.7 mL will be taken at one time, i.e. 27 mL per patient..
  The tubes will be added to the usual blood sample taken at the same time as the patient's usual follow-up consultation.
  To meet the various objectives, we will analyse this blood as follows:
  * Analysis of platelet-poor plasma
  * Analysis of platelet-rich plasma
  * Thrombin generation test with Mim8 and other triggers
  * Electron microscopy (SEM) analysis of the blood clots obtained
  * Analysis of viscoelasticity using ROTEM®.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adults patients with severe hemophilia A (FVIII<2%): Adults patients with severe hemophilia A (FVIII<2%) who are:
  * on prophylaxis with FVIII concentrates after a washout period of 48h for SHL FVIII molecules and at least 4 days for EHL FVIII
  * or receive on demand FVIII treatment without any FVIII treatment since 48h for SHL FVIII molecules and since 4 days for EHL FVIII
  Interventions: Other: blood test

INTERVENTIONS:
Other: blood test — blood test at the inclusion 10 tubes of 2.7mL blood

SUMMARY:
Hemophilia A is an X linked disorder characterized by a deficiency in Factor VIII. The clinical hallmark of this disease is increased tendency to spontaneous bleeding with hemarthrosis accounting for 90% of the hemorrhages. In addition to development of hemophilic arthropathy, the emergence of alloantibodies that inhibit the coagulant activity of FVIII remains the most feared complication related to the treatment of hemophilia A. 30% of patients with hemophilia A develop these inhibitors, making treatment with standard replacement therapy ineffective. Up until the approval of emicizumab, bypassing agents like activated prothrombin complex concentrate (aPCC) and activated recombinant activated factor VII (rFVIIa) were the only approved therapies for the treatment hemophilia A with inhibitors. The response to bypassing therapy is often unpredictable, variable and difficult to monitor.

Emicizumab is a first generation bispecific antibody mimicking the activity of FVIIIa in tenase complex. Early in the HAVEN 1 clinical trial with emicizumab (1), cases of thrombotic microangiopathy (TMA) and thrombotic events were reported when on average a cumulative amount of >100 U/kg/24 hours of aPCC was administered for 24 hours or more to patients receiving emicizumab, resulting in a protocol adjustment for the HAVEN 1 trial and subsequent trials to recommend using the lowest doses of bypassing agents expected to achieve hemostasis, and avoiding the combination of emicizumab and aPCC if possible. So far the only proposed strategies for treating events of breakthrough bleeds in patients on emicizumab prophylaxis include rFVIIa, FVIII in patients with a low titer of inhibitors, and lower doses of aPCC, knowing that emicizumab provides an existing level of thrombin generation. (2) While the exact mechanism leading to the development of thrombotic complications (TMA and VTE) remains poorly understood, many speculated on the accumulation of FIX and FX, the substrates of emicizumab, with multiple doses of aPCC (3)

Mim8 is a novel, next-generation FVIIIa mimetic designed for the subcutaneous prophylactic treatment of patients with HA with and without inhibitors. Mim8 is a fully human, bispecific antibody that mimics FVIIIa function by bridging FIXa and FX on the phospholipid surface of activated platelets, enhancing the proteolytic activity of FIXa, and thus facilitating effective FX activation. Data from studies using in vitro HA-like human blood, as well as in vivo HA mouse models, indicate that Mim8 is ~15-fold more potent than a sequence identical analogue (SIA) of the FVIII mimetic emicizumab (4). Mim8 nonclinical safety program in cynomolgus monkeys showed that subcutaneous administration of up to 3 mg/kg/week (several fold greater than expected clinical exposure) for 26 weeks resulted in relevant pharmacodynamic effects, observed in thrombin generation and APTT, with no signs of thrombi or excessive coagulation activation. So far, Mim8 procoagulant activity was evaluated in platelet poor plasma samples only (5,6)

This in vitro study aims to evaluate TGA to monitor Mim8. We hypothesized that TG profiles (ETP and peak thrombin) may be different with different triggers used. We recently modified TGA to better detect haemostatic activity of emicizumab, by using a combined trigger (low TF+low FIXa). Differently from emicizumab, Mim8 stimulates the proteolytic activity of FIXa in the range of 15,000-fold. TGA test conditions may be therefore different for Mim8 and emicizumab.

ELIGIBILITY:
Inclusion Criteria:

* Male patients,
* Age > 18 years at time of inclusion
* Diagnosis of severe hemophilia A (FVIII <2%)
* Severe hemophilia A (FVIII <2%) and not receiving emicizumab prophylaxis
* Obtaining the patient's non-opposition
* Ability to comply with the study protocol, in the investigator's judgment

Exclusion Criteria:

* Not willing to provide extra blood for the experiments
* Patients carrying the diagnoses of other coagulopathies in addition to hemophilia A
* Patients that have received any hemostatic agent within 5 half-lives of the blood draw.

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 6 Adults patients with severe hemophilia A (FVIII<2%) who are:
  * on prophylaxis with FVIII concentrates after a washout period of 48h for SHL FVIII molecules and at least 4 days for EHL FVIII
  * or receive on demand FVIII treatment without any FVIII treatment since 48h for SHL FVIII molecules and since 4 days for EHL FVIII
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2024-03-28 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
Determination of thrombin generation (TG) (ETP and peak thrombin) will be obtained in platelet-poor plasma from patients with severe HA | One point at the inclusion
  27 ml blood samples will be taken from each patient, and FVIII activity will be measured in the samples. Mim8 and emicizumab will be added to the blood samples, and thrombin generation will be performed using different triggers.
  All statistical analyses were performed using GraphPad Prism and GraphPad Instat softwares (GraphPad Software, La Jolla, CA, USA). The probability of statistical difference between experimental groups will be determined by unpaired Mann-Whitney and ANOVA tests. Results will be expressed as mean ± standard deviation (SD). A p-value < 0.05 will be considered statistically significant

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Référence Hémophilie, Hôpital Louis Pradel- Hospices Civils de Lyon, Bron, Rhone, France

IPD SHARING:
Plan to Share IPD: No